CLINICAL TRIAL: NCT00096707
Title: Phase I Dose Escalation Trial of 2-Deoxy-D-Glucose (2DG) Alone and in Combination With Docetaxel in Subjects With Advanced Solid Malignancies
Brief Title: Dose Escalation Trial of 2-Deoxy-D-Glucose (2DG) in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Threshold Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-101
Record Dates: First submitted 2004-11-12; First posted 2004-11-15 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Lung Cancer; Breast Cancer; Pancreatic Cancer; Head and Neck Cancer; Gastric Cancer
Keywords: advanced solid tumors; cancer; docetaxel; 2-deoxy-D-glucose (2DG); phase 1
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Head and Neck Neoplasms; Stomach Neoplasms; Neoplasms | interventions — Deoxyglucose

INTERVENTIONS:
Drug: 2-deoxy-D-glucose (2DG)

SUMMARY:
The objectives of this study are to evaluate the safety, tolerability, pharmacokinetics, and biologic effect (FDG PET, preliminary efficacy) of daily oral doses of 2DG with and without weekly docetaxel in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
2-deoxy-D-glucose (2DG) is a synthetic glucose analog under development by Threshold Pharmaceuticals, Inc. that exploits the differences in metabolism between normal and malignant cells. Malignant cells utilize glucose at a much higher rate than normal cells and are therefore more dependent on aerobic and anaerobic glycolysis. If glycolysis could be blocked preferentially in malignant cells, 2DG would have potential for anti-tumor therapy. Hypoxic cells are especially dependent on anaerobic glycolysis and are generally resistant to anti-tumor therapies such as chemotherapy and radiotherapy. Therefore, combining 2DG with chemotherapy may be a way to simultaneously target both hypoxic and aerobic cells in tumors.

Four factors may play a role in the preferential toxicity of 2DG in malignant cells: (1) increased uptake and retention of glucose analogs by malignant cells; (2) relative hypoxia of tumor cells relative to normal cells; (3) malignant cells may be more sensitive to glucose deprivation than normal cells; and (4) inhibition of glycolysis may increase sensitivity to some cytotoxic agents. Preliminary data in human tumor xenografts support this hypothesis.

Because 2DG is most likely to be effective in combination with chemotherapy, this trial was designed to evaluate the maximum tolerated dose (MTD) of 2DG both alone and in combination with chemotherapy. Docetaxel was chosen because there is evidence in human tumor xenografts of delayed tumor growth for 2DG in combination with paclitaxel compared to paclitaxel alone and it has been reported that taxanes may enhance uptake of 2DG into malignant cells. Patients with advanced solid tumors were chosen because they are appropriate candidates for a Phase I clinical trial and because their tumors are likely to have areas of hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, at least 18 years of age
* Histologically confirmed, locally advanced or metastatic solid malignancy
* Previously treated with at least one chemotherapy regimen for advanced or metastatic disease OR no curative standard treatment is available
* Recovered from reversible toxicities of prior therapy
* Life expectancy of at least 3 months
* ECOG performance status of 0, 1, or 2
* Measurable or nonmeasurable disease by RECIST criteria
* Ability to understand the purposes and risks of the study and having signed a written informed consent form
* All women of childbearing potential and all men must agree to use effective means of contraception from entry into the study through 3 months after the last dose

Exclusion Criteria:

* Previous or current CNS metastases (screening CT or MRI is not required in asymptomatic subjects)
* Active clinically significant infection requiring antibiotics
* Known glucose-6-phosphate dehydrogenase deficiency or history of anemia of unknown etiology
* History of clinically significant unexplained episodes of hypotension, fainting, dizziness, or lightheadedness
* History or symptoms of cardiovascular disease, particularly coronary artery disease, arrhythmias, or conduction defects with risk of cardiovascular instability, uncontrolled hypertension, clinically significant pericardial effusion, or congestive heart failure
* History of transient ischemic attack, stroke, or seizure disorder or any other CNS disease considered to be significant by the investigator
* Known autonomic dysfunction or chronic orthostatic hypotension
* Evidence of hypoglycemia, clinically significant renal disease, clinically significant liver disease (other than liver metastases), diabetes mellitus, gastrointestinal disorder (that could affect absorption or elimination of orally-administered medications), or obstructive uropathy with significant post-void residual during the past 5 years
* Known HIV infection
* Other primary malignancies (other than treated basal cell carcinoma of the skin or treated in situ cervical cancer) within the past 5 years
* Major surgery within 4 weeks of the start of study treatment, without complete recovery
* Antitumor therapy within 21 days of the start of study treatment
* Disease progression/relapse on docetaxel therapy within the past 12 months
* A history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* Known sensitivity to methylparaben or propylparaben
* Inability to discontinue prohibited medications for 24 hours before and after dosing on Day 1 of Weeks 1, 2, and 3 and Day 5 of Week 1. In addition, patients who cannot discontinue medications known to induce or inhibit CYP 3A4, such as cyclosporine, terfenadine, ketoconazole, erythromycin, and troleandomycin, for the duration of the study are not eligible.
* Peripheral neuropathy >= Grade 2
* Hemoglobin <9 g/dL
* ANC <1500/μL
* Platelet count <100,000/μL
* Total bilirubin >1.5 mg/dL
* Abnormal liver function
* Serum creatinine >1.5 mg/dL unless creatinine clearance is >= 60 mL/min
* Serum potassium < lower limit of normal
* Elevated fasting blood glucose
* Pregnant or nursing women
* Participation in an investigational drug or device study within 28 days of the first day of dosing on this study
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study.
* Unwillingness or inability to comply with the study protocol for any other reason
* Subjects who live alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Significant Toxicity
Disease Progression

SECONDARY OUTCOMES:
Response Rate
Death

CONTACTS AND LOCATIONS:
Overall Officials: Luis Raez, MD, Principal Investigator — University of Miami Sylvester Comprehensive Cancer Center
Locations (3):
- United States (3):
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Institute for Drug Development Cancer Therapy & Research Center, San Antonio, Texas

REFERENCES:
- [Derived] Raez LE, Papadopoulos K, Ricart AD, Chiorean EG, Dipaola RS, Stein MN, Rocha Lima CM, Schlesselman JJ, Tolba K, Langmuir VK, Kroll S, Jung DT, Kurtoglu M, Rosenblatt J, Lampidis TJ. A phase I dose-escalation trial of 2-deoxy-D-glucose alone or combined with docetaxel in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2013 Feb;71(2):523-30. doi: 10.1007/s00280-012-2045-1. Epub 2012 Dec 11. PMID 23228990
- See also: Threshold Pharmaceuticals Homepage — http://www.thresholdpharm.com